CLINICAL TRIAL: NCT06992219
Title: Effects of Minimally Non-surgical Periodontal Treatment Versus Quadrantwise Subgingival Instrumentations on Infrabony Defects and Analysis of Defect Morphology on the Effectiveness of Treatment
Brief Title: Impact of Minimally Invasive Non-surgical Periodontal Treatment on Infrabony Defects
Acronym: Infra-MINST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-3308
Record Dates: First submitted 2025-05-18; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Intrabony Defect
Keywords: periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Non-surgical periodontal treatment Subgingival biofilm ultrasonic debridement with MINST or Q-SI for infrabony defects
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST non surgical periodontal treatment (Experimental): MINST non surgical periodontal treatment Periodontitis patients treated by means of MINST for infrabony defects. Patients were treated with non-surgical MINST periodontal treatment in a single session.
  Interventions: Other: Non surgical periodontal treatment evaluated through probing pocket depth reduction
- Q-SI non surgical periodontal treatment (Active Comparator): Periodontitis patients treated by means of Q-SI. Patients were treated with non-surgical quadrantwise periodontal treatment in 4 sessions, 1 session per week.
  Interventions: Other: Non surgical periodontal treatment evaluated through probing pocket depth reduction

INTERVENTIONS:
Other: Non surgical periodontal treatment evaluated through probing pocket depth reduction — Patients were treated with Minimally invasive non surgical treatment (MINST) or quadrant-subgingival instrumentation (Q-SI). The efficacy of treatment in both groups was evaluated through Probin Pocket Depth reduction in millimetres measurement before and after treatment.

SUMMARY:
Fifty-two periodontitis patients (26 per group) were randomly assigned to the test (Minimally invasive non-surgical therapy - MINST) or the control group (Quadrantwise Subgingival Instrumentation - Q-SI) NPT protocols.

DETAILED DESCRIPTION:
Clinical periodontal parameters, the number of pocket sites, x-ray of the infrabony defects characteristics and a composite outcome measure (COM) on the combined assessment of intrabony defect were recorded at baseline, and -3, 6- and at 12-months after treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Periodontitis

Exclusion Criteria:

* Periodontal treatment
* Use of antibiotics, NSAIDs, and immunosuppressants during the last 6 months
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth Reduction | 1-year
  Probing Pocket Depth Reduction in Probing Pocket Depth after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, DDS, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Study results